CLINICAL TRIAL: NCT06709872
Title: Discriminating Borderline from Stage I Invasive Ovarian Cancer (BIOC): a Prospective Multicenter Diagnostic Biomarker Study
Brief Title: A Prospective Multicenter Diagnostic Biomarker Study to Discriminate Borderline from Stage I Invasive Ovarian Cancer
Acronym: BIOC
Status: Active, not recruiting | Type: Observational
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, An Coosemans, Head of the Laboratory at KU Leuven and Gynaecologist (Dr. Prof.), KU Leuven
Other Study IDs: S69849; 13583 (Other Grant/Funding Number: Stand up to Cancer (Kom op tegen Kanker))
Record Dates: First submitted 2024-11-26; First posted 2024-11-29 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Stage I Ovarian Cancer; Borderline Ovarian Tumors
Keywords: Borderline ovarian tumors; stage I ovarian cancer; diagnostic; biomarkers
MeSH Terms: conditions — Ovarian Neoplasms; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Serum isolated from blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Borderline ovarian tumor cohort: Patients with ultrasound discovery of a cyst on the ovary, suspicious for BOT
- stage I invasive ovarian cancer cohort: Patients with ultrasound discovery of a cyst on the ovary, suspicious for stage I invasive ovarian cancer

SUMMARY:
The study aims to improve the diagnosis of ovarian cancer by distinguishing between borderline ovarian tumors (BOT) and stage I invasive ovarian cancer. Other than the traditional diagnostic biomarker CA125, the previous study TRANS-IOTA (translational-international ovarian tumor analysis; S51375/S59207), conducted by similar investigators, pointed at biomarkers like HE4, CA72.4, CA15.3, and CCL11, as potential markers to discriminate BOT from stage I cancer. BIOC is the follow-up study, which will include four additional promising biomarkers to expand the panel to nine. The investigators aim to confirm whether a subpanel of these nine biomarkers has diagnostic value. Such a biomarker signature would enhance the accuracy of distinguishing between BOT and stage I invasive ovarian cancer before surgery, leading to more precise treatment and improved patient outcomes.

DETAILED DESCRIPTION:
The BIOC study, titled Discriminating Borderline from Stage I Invasive Ovarian Cancer, is a prospective, multicenter diagnostic biomarker study designed to refine diagnostic accuracy for ovarian cancer, specifically to differentiate between borderline ovarian tumors (BOT) and stage I invasive ovarian cancer. Existing diagnostic tools, such as the CA125 biomarker, are limited in their ability to provide precise differentiation in early stages, which is crucial for appropriate pre-surgical treatment planning. This study builds upon findings from the TRANS-IOTA (translational-international ovarian tumor analysis) study, expanding the biomarker panel to nine proteins, including CA125, HE4, CA72.4, and CCL11, alongside four additional biomarkers selected through systematic literature review.

The primary objective of BIOC is to develop a biomarker signature capable of distinguishing BOT from early-stage invasive ovarian cancer. This would allow for more accurate diagnoses either independently or in combination with ultrasound variables, thereby improving pre-surgical decision-making, reducing the need for second surgeries, and supporting more tailored treatments that improve patient outcomes. For younger patients with BOT, for instance, accurate differentiation could allow for fertility-preserving surgical options. A secondary aim of the study is to establish a robust database for BOT and stage I invasive ovarian cancer across Flanders (Belgium) and Europe, capturing detailed clinical, ultrasound, histological, and immune data that will guide future research and support gynecologists in refining their diagnostic approaches.

BIOC will be conducted across multiple hospitals in Flanders (Belgium) and a few European centers and aims to enroll 200 patients with BOT and 200 with stage I invasive ovarian cancer. Participants will primarily be recruited through gynecology ultrasound departments, where they will receive pre-surgical blood sampling and clinical evaluations. Recruitment will occur over three years, with the study concluding after a subsequent two-year analysis period, aiming for completion between 2028 and 2029.

By establishing a validated biomarker panel for early ovarian cancer diagnosis, BIOC has the potential to significantly enhance diagnostic accuracy and efficiency. This could transform the precision of preoperative assessments, reduce unnecessary invasive procedures, and improve overall treatment planning, thus enhancing patient outcomes and quality of life for those affected by ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Participants eligible for inclusion in this study must meet all of the following criteria:

  1. Voluntary written informed consent of the participant or their legally authorized representative has been obtained prior to any screening procedures
  2. At least 18 years of age at the time of signing the Informed Consent Form (ICF)
  3. Ultrasound discovery of a cyst on the ovary, suspicious for BOT or stage I invasive tumor (subjective assessment)

Exclusion Criteria:

* Participants eligible for this Study must not meet any of the following criteria:

  1. Participants younger than 18 years old,
  2. Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using an adequate, highly effective contraceptive
  3. Participants who refuse the preoperative transvaginal ultrasonography and/or blood sample
  4. Participants with known simultaneous and/or previous malignancies within five years prior to BIOC participation
  5. Participants with infectious serology (i.e. HIV, Hepatitis B, Hepatitis C)
  6. Participants who deny or withdraw the written informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — All females with female reproductive system as this study aims to improve diagnosis of ovarian cancer
Study Population: Patients with ultrasound discovery of a cyst on the ovary, suspicious for BOT or stage I invasive tumor
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-09-03 (Actual); Primary Completion 2029-09-03 (Estimated); Study Completion 2029-09-03 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of biomarkers | After 12 months following the recruitment
  Diagnostic performance of a protein-based biomarker or set of biomarkers that can discriminate between BOT and stage I invasive ovarian cancer in terms of area under the receiver operative characteristics curve (AUROC).

SECONDARY OUTCOMES:
Database establishment | Start registering the data of patients in the database from the day of recruitment
  Establishment of a database for borderline ovarian tumors (BOT) and stage I invasive ovarian cancer to address future research questions.

CONTACTS AND LOCATIONS:
Overall Officials: An Coosemans, Principal Investigator — KU Leuven
Locations (1):
- UZ Leuven, Leuven, Flemish Brabant, Belgium